CLINICAL TRIAL: NCT05545748
Title: The Effect of a Zero Tolerance Program (SToP) Applied to Parents of Children at High Risk of Secondhand Tobacco Smoke Exposure on Child's Urine Cotinine Level According to Exposure Feedback: A Randomized Controlled Study
Brief Title: The Effect of a Zero Tolerance Program (SToP) on Child's Urine Cotinine Level According to Exposure Feedback
Acronym: SToP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Sebahat Gozum, Prof.Dr.Sebahat Gozum, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0015
Record Dates: First submitted 2022-09-12; First posted 2022-09-19 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Second Hand Smoke; Exposure to Environmental Pollution; Child; Urine; Parents
Keywords: Urinary cotinine; Home environment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participating parents will not know which group they are. Also, when the data is analyzed by the statistician, she/he will not know which group it is.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zero (0) Tolerance Program Group (Experimental): The intervention to this group consists of four parts.
  1. Urine Cotinine Feedback: Explaining what the cotinine-sensitive dipstick test kit score and color scale mean. Cotinine-sensitive dipstick test kit is a simple, cost-effective test to determine smoking status. It is an easy-to-read test strip that can be used with either a saliva or a urine sample.
  2. Giving reminder objects (Magnet, sticker): For example; at the entrance door of the house: "0 TOLERANCE" magnet to cigarettes; "No smoking in my home" label.
  3. Informative Materials (Information Notes and Brochures): Brochures on the harms of second-hand smoking (SHS) and third-hand smoking (THS), the diseases they cause, and how to protect them
  4. Informative Telephone Text Messages: Reminder phone messages related to SHS and THS
  Interventions: Behavioral: Zero (0) Tolerance Program (SToP)
- Exposure Feedback Group (Active Comparator): This group will receive only exposure feedback Urine Cotinine Feedback: Explaining what the cotinine-sensitive dipstick test kit score and color scale mean. Cotinine-sensitive dipstick test kit is a simple, cost-effective test to determine smoking status. It is an easy-to-read test strip that can be used with either a saliva or a urine sample.
  Interventions: Behavioral: Exposure Feedback Group

INTERVENTIONS:
Behavioral: Zero (0) Tolerance Program (SToP) — 1. Urine Cotinine Feedback: Explaining what the cotinine-sensitive dipstick test kit score mean. Cotinine-sensitive dipstick test kit is a simple, cost-effective test to determine smoking status. It is an easy-to-read test strip that can be used with either a saliva or a urine sample.
  2. Giving reminder objects (Magnet, sticker): For example; at the entrance door of the house: "0 TOLERANCE" magnet to cigarettes; "No smoking in my home" label.
  3. Informative materials (information notes and brochures): Brochures on the harms of second-hand smoking (SHS) and third-hand smoking (THS), the diseases they cause, and how to protect them
  4. Informative telephone text messages: Reminder phone messages related to SHS and THS
  Arms: Zero (0) Tolerance Program Group
Behavioral: Exposure Feedback Group — 1. Urine Cotinine Feedback: Explaining what the cotinine-sensitive dipstick test kit score mean. Cotinine-sensitive dipstick test kit is a simple, cost-effective test to determine smoking status. It is an easy-to-read test strip that can be used with either a saliva or a urine sample.
  Arms: Exposure Feedback Group

SUMMARY:
Although the ban on indoor smoking has greatly reduced secondhand smoke (SHS) exposure in public spaces, the home environment is still the primary source of exposure to SHS, particularly in children under the age of five. Although attempts are often made to prevent or reduce children's exposure to SHS, such as education, counseling, and exposure feedback to parents, exposure remains. Although using materials such as brochures, messages, posters and reminders that will minimize the harms such as protecting children from SHS will reduce the exposure, exposure continues in the long term.The aim of this study is to compare the effect of giving exposure feedback to the parents according to the zero tolerance program (SToP) on the urinary cotinine level of the children. In this study with active control group, single-blind (participant), randomized control, stratified block randomization (1:1) will be performed. Totally 58 participants including STOP intervention group (n:29) and the exposure feedback group (n:29), which is the active control group, were planned to be included in the study, which was planned to be conducted between January and September 2023. Cotinine-sensitive dipstick test kits will be used for the primary outcome (urine cotinine). Cotinine-sensitive dipstick test kit is a simple, cost-effective test to determine smoking status. It is an easy-to-read test strip that can be used with either a saliva or a urine sample. Secondary outcomes will be evaluated by information form on exposure to second-hand smoke, an attitude form on exposure to second-hand smoke, and a scale of beliefs towards third-hand smoke. This protocol will demonstrate whether SToP interventions, a sustainable program for children at high risk of secondhand tobacco exposure, are a viable intervention for parents on how to reduce exposure.

ELIGIBILITY:
Inclusion Criteria:

* Parents with children aged 5 and under, whose children are registered with the Family Health Center, and whose children are at high and very high risk of exposure to SHS according to the risk algorithm.
* Parents' willingness to participate in the study

Exclusion Criteria:

* Babysitter
* Those who do not speak Turkish.
* Parents of children with asthma will not be included on the grounds that it may be confusing as they may display more specific behavior.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2023-12-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Urine Cotinine Level | Change in Urine Cotinine Level at 3 and 6 months from baseline
  The child's urine sample taken at any time will be analyzed with the cotinine-sensitive dipstick test kit to assess the urine cotinine level. Urine samples will be tested in accordance with the manufacturer's instructions. The test has over 99% sensitivity in detecting cotinine with a cut-off level of 200 ng/ml and a minimum detection time of 2-8 hours and a maximum detection time of 1-7 days. After the test is immersed in the urine collection container for 10 seconds, the result becomes clear within 5 minutes. If the test is negative, the control (C) and test (T) line appear. If the test is positive, only the control line (C) appears. If the C and T lines are not visible or the C line is visible, it means that the test is invalid. Each test sample will be read and recorded by two independent observers.

SECONDARY OUTCOMES:
The Information Form on Exposure to Secondhand Smoke | Change in knowledge level at 3 and 6 months from baseline
  The information form created by the researchers consists of 16 items: for each item; right, wrong, I don't know, can choose one of the options. Each item is scored between 0 and 1 according to the answer given. Accordingly, scores ranging from 0-13 for the first section, 0-3 for the second section, and 0-16 for the sum of the information items are taken. An increase in the score is interpreted as good knowledge of SHS and THS. The Kuder Richardson 20 (KR-20) value of all items was found to be 0.84.
Attitude Form on Exposure to Secondhand and Third hand Smoking | Change in attitude level at 3 and 6 months from baseline
  There are 8 attitude statements in the Household Attitude Form on Exposure of Children Under Five to Secondhand Smoking. 1 point for positive attitude statements and 0 (zero) points for negative attitude statements. Accordingly, the attitude score for exposure to second-hand smoking can be taken between 0-6, the tobacco attitude score for third-hand exposure 0-2, and the total attitude score to 0-8. A high score indicates a positive attitude.The KR-20 value of the expressions related to second-hand smoking exposure was found to be 0.84, the Kuder Richardson 20 (KR-20) value of the expressions related to the third-hand smoking exposure was found to be 0.53 and the KR-20 value of the total attitude expressions was 0.77.
Beliefs About Third-Hand Smoke (THS) Scale | Change in beliefs level at 3 and 6 months from baseline
  The scale, which consists of nine items, is answered in a 5-point Likert type. The scale was developed in United States in 2017 to determine beliefs about Third-Hand Smoke (THS). The Turkish validity and reliability study of the scale was carried out in 2019. As the score from the scale gets closer to 5, it is interpreted that the individual believes in the effects of THS on the environment and health, and as it approaches 1, the individual does not believe in the effects of THS on the environment and health.

CONTACTS AND LOCATIONS:
Locations (1):
- Sebahat Gözüm, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No